CLINICAL TRIAL: NCT02714543
Title: Evaluation of Efficacy of Aloevera in the Treatment of Oral Submucous Fibrosis- A Clinical Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Oxford Dental College, Hospital and Research Center, Bangalore, India (Other)
Responsible Party: Principal Investigator, Dr. Anuradha Pai, Professor and Head, Dept of oral medicine and radiology, The Oxford Dental College, Hospital and Research Center, Bangalore, India
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OxfordDC
Record Dates: First submitted 2016-02-19; First posted 2016-03-21 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-03

CONDITIONS: Oral SubMucous Fibrosis
Keywords: OSMF; Aloevera; Hydrocortisone; Hyaluronidase
MeSH Terms: conditions — Oral Submucous Fibrosis | interventions — Hydrocortisone; Hyaluronic Acid; Antioxidants

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- aloevera group (Experimental): aloevera juice twice daily for 3 months. aloevera gel one scoop to be applied 3-4 times daily for 3 months
  Interventions: Drug: aloevera juice; Drug: aloevera gel
- steroid group (Active Comparator): intralesional injection of hydrocortisone 100mg and injection hyaluronic acid 1500IU once a week for 6 weeks with Capsules SM Fibro once daily for 3 months.
  Interventions: Drug: Hydrocortisone; Drug: Hyaluronic Acid; Drug: antioxidant

INTERVENTIONS:
Drug: aloevera juice — aloevera juice to drink twice daily for 3 months.
  Arms: aloevera group
Drug: Hydrocortisone — intralesional injection of hydrocortisone 100mg once a week for 6 weeks
  Arms: steroid group
Drug: Hyaluronic Acid — injection hyaluronic acid 1500IU once a week for 6 weeks
  Arms: steroid group
Drug: antioxidant — Capsules SM Fibro (antioxidants) once daily for 3 months.
  Other Names: Capsule SM Fibro
  Arms: steroid group
Drug: aloevera gel — aloevera gel one scoop to be applied 3-4 times daily for 3 months
  Arms: aloevera group

SUMMARY:
Oral submucous fibrosis is a chronic, insidious disease caused by arecanut use and is associated with both significant morbidity (including burning sensation and reduced oral opening) and an increased risk of malignancy. Treatment of Oral SubMucous Fibrosis has largely been symptomatic and is associated with high recurrence rate. Aloevera has immunomodulatory, anti-inflammatory, wound healing, antioxidant and antineoplastic activities. All such properties of Aloevera suggest the possibility of its use in the management of oral submucous fibrosis.

In the present study, 74 patients of Oral SubMucous Fibrosis were randomly divided into 2 groups (Group A & B). Group A patients were instructed to drink 30ml of aloe vera juice twice daily before food and to apply 5mg (approx 1 scoop) of aloe vera gel over the lesion 3-4 times daily for 3 months. Group B patients were given intralesional injections of 1.5ml Hydrocortisone acetate 25mg/ml and hyaluronidase (1500 IU) weekly for 6 weeks. They were also prescribed SM Fibro (Alpha lipoic acid 50mg, Beta-carotene 10mg, Elemental copper 1mg, Elemental selenium 75mcg, Lycopene 5mg, Vitamin E 10 IU, Zinc sulphate 27.45mg in form of the capsule) for 3 months. Patients were assessed for burning sensation, interincisal mouthopening, cheek flexibility and tongue protrusion at an interval of 1, 2 and 3 months.

DETAILED DESCRIPTION:
Material and Methods The present study was conducted in the Department of Oral Medicine and Radiology at The Oxford Dental College and Hospital, Bangalore, India between November 2013 to August 2015. Approval from the institutional ethical committee was obtained for the study. Patients with Oral SubMucous Fibrosis (Stage 2 according to Pindborg) were enrolled in the study. Pregnant women, lactating mothers, patients with known history of hypersensitivity to aloevera and those who had received prior treatment for OSMF were excluded. 74 patients who were ready to quit the habit and accept regular follow up treatment protocol were included in the study. An informed consent was obtained from all the patients after the nature of the study and its procedures were explained. A thorough clinical examination was done and the following parameters were measured and recorded by an independent examiner.

1. The intensity of burning sensation was recorded using a Numerical Rating Visual Analogue Scale.
2. The interincisal mouth opening was measured using a metal scale and divider from the mesioincisal angle of upper central incisor to the mesioincisal angle of lower central incisor and recorded in millimeters.
3. Cheek flexibility (CF) was measured according to the method described by Bailoor and Nagesh. Two points were marked, one on each side of the face at 1/3rd the distance from angle of the mouth on a line joining the tragus of the ear and the angle of the mouth. The distance measured between these two points was V2. The subject was asked to blow his cheek fully and the distance measured between the same two points was V1. CF=V2-V1.
4. Tongue protrusion was assessed from normal mesioincisal angle of upper central incisor to the tip of the tongue when maximally extended with mouth wide open.

The patients were randomly divided into 2 groups (Group A & B). Group A patients were given pure aloevera gel and pure aloevera juice (Processed and manufactured by Hemant Sai, Sun Vision Company, Neel RLI Pvt Ltd). They were instructed to drink 30ml of aloevera juice twice daily before food and to apply 5mg (approx 1 scoop) of aloevera gel over the lesion 3 times per day for 3 months. Group B patients were given intralesional injections of Hydrocortisone acetate 25mg/ml and hyaluronidase (1500 IU) weekly for 6 weeks. They were also prescribed Cap SM Fibro twice daily for 3 months. Same baseline parameters were measured and recorded at an interval of 1, 2 & 3 months by the same examiner who measured the baseline values and was unaware of the treatment received by the study subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically diagnosed stage 2 OSMF patients.
2. Patients who were ready to quit the habit and accept regular follow up protocol.

Exclusion Criteria:

1. Patients with stage 1 & 3 OSMF.
2. Patients with history of hypersensitivity to aloevera.
3. Pregnant women & lactating mothers.
4. Patients who had undergone any other treatment for OSMF.

Ages: 17 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 74 (Actual)
Dates: Start 2013-11; Primary Completion 2015-08 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
burning sensation | 3 months
  Visual analogue scale
mouth opening | 3 months
  interincisal mouth opening was measured using a metal scale and divider from the mesioincisal angle of upper central incisor to the mesioincisal angle of lower central incisor and recorded in millimeters
cheek flexibility | 3 months
  Two points were marked, one on each side of the face at 1/3rd the distance from angle of the mouth on a line joining the tragus of the ear and the angle of the mouth. The distance measured between these two points was V2. The subject was asked to blow his cheek fully and the distance measured between the same two points was V1. CF=V2-V1. measured in milimeters
tongue protrusion | 3 months
  from mesioincisal angle of upper central incisor to the tip of the tongue when maximally extended with mouth wide open. measured in milimeters